CLINICAL TRIAL: NCT05271669
Title: Patterns of SARS-CoV-2 Immunity At Household Level and Their Changes Over Time
Brief Title: COVID-19 Immunity and Changes Over Time
Status: Withdrawn | Type: Observational
Why Stopped: Changes in COVID-19 situation with repeated shut-down making it imposible to enrol subjects during 2022
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shui-Shan Lee, MD, Research Professor, Chinese University of Hong Kong
Other Study IDs: Protocol HK COVID cohort 2021
Record Dates: First submitted 2022-03-07; First posted 2022-03-09 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
Keywords: serology; cohort study; SARS-CoV-2 antibody
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for serology testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The risk of household spread of SARS-CoV-2 hinges on both the transmission dynamics of the virus circulating in the community as well as the seroprotection pattern of constituent members, which can be attributed to vaccination and previous infections. This study is conceptualised to assess the dynamicity of SARS-CoV-2 risk at the household level, through monitoring the pattern of seroprotection, in conjunction with the vaccination coverage, history of infection and exposure risk in the setting of Hong Kong.

DETAILED DESCRIPTION:
The aim of this study is to assess the SARS-CoV-2 risk at the household level, with the objectives of (a) determining the coverage of vaccination and its changes over time; (b) monitoring pattern of exposure and history of infection; and (c) evaluating the level of seroprotection and its longitudinal trend.

A cohort of households comprising 900 persons would be recruited. Invited participants would be attend the Research Centre for blood sampling and the completion of a simple questionnaire at 3 different timepoints at 12-18 months apart. A questionnaire would be administered to capture the following characteristics: (a) Socio-demographics; (b) History of SARS-CoV-2 infection; (c) adoption of precautionary measures; (d) SARS-CoV-2 testing history and (e) SARS-CoV-2 vaccination uptake.

Participants would be tested for SARS-CoV-2 serology. The main markers for measurement are nucleocapsid antibody for inferring past infection, spike antibody for the immunological responses, and seroprotection by SARS-CoV-2 surrogate virus neutralisation test.

ELIGIBILITY:
Inclusion Criteria:

* adults of age 18 or above, or children under the age of 18 with informed consent of the legal guardian
* normally residing in Hong Kong
* could communicate in spoken and written Chinese and/or English

Exclusion Criteria:

* individuals with mental illness
* prisoners

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults of households enrolling in a population cohort covering residents from all 18 districts in Hong Kong.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with COVID-19 protective immunity | 1 year
  Prevalence of SARS-CoV-2 spike antibody
Proportion of participants with marker of past COVID-19 infection | 1 year
  Prevalence of SARS-CoV-2 nucleocapsid antibody

CONTACTS AND LOCATIONS:
Locations (1):
- Shui Shan Lee, Hong Kong, HONG KONG, China